CLINICAL TRIAL: NCT04832217
Title: Innovaciones Aplicadas a la Cadena Productiva Pirenaica de Vacuno Para Valorizar Una Carne Identificable Por el Consumidor.
Brief Title: Innovations Applied to the Pyrenean Beef Production to Enhance Consumer-identifiable Meat.
Acronym: DIETAPYR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Luis Alberto Moreno Aznar, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EFA 144/16
Record Dates: First submitted 2021-03-24; First posted 2021-04-05 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Body Weight Changes; Habits, Diet; Habit, Food; Life Change Events
Keywords: randomized controlled crossover trial; young adults; Pyrenean beef
MeSH Terms: conditions — Body Weight Changes; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: A cross-over randomized controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pyrenees' beef group (Experimental): In the first period, 24 participants were randomly assigned to a beef (Pyrenees' beef group).
  In the second period, 23 participants were randomly assigned to a beef (Pyrenees' beef group).
  Interventions: Other: Pyrenees´ Beef diet
- Conventional Chicken group (No Intervention): In the first period, 23 participants were randomly assigned to a conventional chicken-based group (control group).
  In the second period, 24 participants were randomly assigned to a conventional chicken-based group (control group).

INTERVENTIONS:
Other: Pyrenees´ Beef diet — 24 participants were randomly assigned to a Pyrenees' beef diet, 3 serving per week during of 8 weeks.
  Arms: Pyrenees' beef group

SUMMARY:
The DIETAPYR2 study is a randomized controlled crossover trial consisting of two experimental periods each lasting 8 weeks. Enrolled participants were randomly assigned to either a Pyrenean beef-based diet or a conventional chicken-based diet and instructed to consume this meat three times a week.

In the first visit the medical history was obtained and anthropometric measurements, blood pressure (systolic and diastolic) and heart rate were taken. The day after the first visit, in the morning, a sample of blood, stool and urine was taken from the participants after an overnight fast. At the time of this visit (period 1), each participant was randomly assigned to a Pyrenean beef diet (intervention group) or a conventional chicken-based diet (control group).

After an experimental period of 8 weeks, the participants were invited to carry out the same evaluations as during the first visit. Subsequently, a 5-week washout period was carried out to eliminate the possible residual effects of the first experimental period. After the washout period, the participants were called back for the same assessments during a third visit just before the second experimental period (period 2). During this period, those who were previously on a Pyrenean beef diet (intervention group) were crossed with the conventional chicken diet (control group) and vice versa. Finally, after the second 8-week experimental period, the participants were retested as on previous visits.

DETAILED DESCRIPTION:
The current study is a sub-study included in the DIETAPYR2 study (Innovations applied to the Pyrenean beef production to enhance consumer-identifiable meat), a randomized-controlled crossover trial consisting of two experimental periods with a duration of 8 weeks each. Enrolled participants were randomly assigned whether to a Pyrenean beef-based diet or to a Conventional chicken-based diet and were instructed to consume this meat three times per week. The Pyrenean beef is meat from young calves of native breeds, raised mainly on local pastures with a recognized impact in environmental and social sustainability of this rural geographical area. The Pyrenees (mountain range between France and Spain) is an optimal place for the practice of extensive livestock rearing given the richness of forages and the existence of native cow breeds that make use of these natural feedstuffs.

To ensure harmonization in the study, each chef of the 3 selected student accommodation halls was provided with instructions on the cooking methods for chicken and beef and they also received examples of recipes. Cooking methods were breaded, stewed and grilled for beef and breaded, stewed and roasted for chicken.

During the 2 weeks before the first period, researchers contacted with participants and obtained informed consent from them. Then, the first visit was scheduled where the medical history was obtained and the anthropometric measurements, blood pressure (systolic and diastolic) and heart rate measures were undertaken. The day after the first visit, in the morning, a blood, stool and urine sample was collected from participants after an overnight fast. At the time of this visit (period 1), each participant was randomly assigned to Pyrenees beef diet (intervention group) or a conventional chicken-based diet (control group).

Following an 8-week experimental period, participants were invited to perform the same assessments as during the first visit. Afterwards, a 5-week washout period took place to remove the possible residual effects of the first experimental period. Participants were requested not to change their diet or physical activity habits for the 5-week washout period. After the washout period, participants were called again to perform the same assessments during a 3rd visit right before the second experimental period (period 2). During this period those previously on Pyrenees beef diet (intervention group) were crossed to conventional chicken diet (control group) and vice versa. Finally, after the 8 week second experimental period, participants were assessed again as in previous visits.

ELIGIBILITY:
Inclusion Criteria:

* To fill a medical history and informed consent to participate.
* Must be able to eat meat and chicken.

Exclusion Criteria:

* Diagnosticated of any chronic, metabolic, endocrine or nutrition related-disease.
* To be vegetarian or vegan
* To be under age (<18 years)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in the triglycerides concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shipped to the laboratory. Standardized laboratory procedures use to analyse samples for triglycerides (mg/dL). Also, the equip VITROS 5600 use to perform the hemogram.
Changes in the HDL cholesterol in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shipped to the laboratory. Standardized laboratory procedures use to analyse samples for high density lipoprotein cholesterol (HDL). Also, the equip VITROS 5600 use to perform the hemogram.
Changes in the LDL cholesterol in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shipped to the laboratory. Standardized laboratory procedures use to analyse samples for low density lipoprotein cholesterol (LDL). Also, the equip VITROS 5600 use to perform the hemogram.

SECONDARY OUTCOMES:
Changes in the iron concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for iron concentration.
  Also, the equip VITROS 5600 use to perform the hemogram.
Changes in the calcium concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for calcium concentration.
  Also, the equip VITROS 5600 use to perform the hemogram.
Changes in the glucose concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for glucose concentration. Also, the equip VITROS 5600 use to perform the hemogram.
Changes in the C-reactive protein in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for C-reactive protein. Also, the equip VITROS 5600 use to perform the hemogram.
Changes in the urea concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for urea concentration. Also, the equip VITROS 5600 use to perform the hemogram.
Changes in the zinc concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for zinc concentration. Also, the equip VITROS 5600 use to perform the hemogram.
Changes in the creatinine concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for creatinine concentration. Also, the equip VITROS 5600 use to perform the hemogram.
Changes in the Palmitic Acid (C16) concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for Palmitic Acid (C16) concentration. Fatty acid will quantified after methylation by gas-liquid chromatography coupled to mass spectrometry detection (GS-MS).
Changes in the Stearic Acid (C18) concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for Stearic Acid (C18) concentration. Fatty acid will quantified after methylation by gas-liquid chromatography coupled to mass spectrometry detection (GS-MS).
Changes in the Oleic Acid (C18_1n9) concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for Oleic Acid (C18_1n9) concentration. Fatty acid will quantified after methylation by gas-liquid chromatography coupled to mass spectrometry detection (GS-MS).
Changes in the Arachidonic Acid (C20_4n6) [AA_W6] concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for Arachidonic Acid (C20_4n6) [AA_W6] concentration. Fatty acid will quantified after methylation by gas-liquid chromatography coupled to mass spectrometry detection (GS-MS).
Changes in the Eicosapentadienoic Acid (C20_5n3) [EPA] concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for Eicosapentadienoic Acid (C20_5n3) [EPA] concentration. Fatty acid will quantified after methylation by gas-liquid chromatography coupled to mass spectrometry detection (GS-MS).
Changes in the Docosahexadienoic Acid (C22_6n3) [DHA] concentration in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Blood sample drew via venipuncture after 12h overnight fast. Sample will immediately shippe to the laboratory. Standardized laboratory procedures use to analyse samples for Docosahexadienoic Acid (C22_6n3) [DHA] concentration. Fatty acid will quantified after methylation by gas-liquid chromatography coupled to mass spectrometry detection (GS-MS).

OTHER OUTCOMES:
Change from baseline in the body fat in those people who Pyrenean beef-based diet compared with the consumption of conventional chicken. | From the beginning of the study to the end of each period of study. 8 weeks per period.
  Body fat percentage will be obtained by the same trained researcher and will be measured with an electronic scale (Tanita BC 418 MA, Tanita Europe GmbH, Sindelfingen, Germany). The participant stand on the platform of the scale without support, with the body weight evenly distributed between both feet. The participant will wear Light indoor clothing, excluding shoes, long trousers and sweater.

CONTACTS AND LOCATIONS:
Locations (1):
- Genud Research Group, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santaliestra-Pasias AM, Miguel-Berges ML, Campo MM, Guerrero A, Olleta JL, Santolaria P, Moreno LA. Effect of the Intake of Lean Red-Meat from Beef-(Pirenaica Breed) versus Lean White-Meat on Body Composition, Fatty Acids Profile and Cardiovascular Risk Indicators: A Randomized Cross-Over Study in Healthy Young Adults. Nutrients. 2022 Sep 9;14(18):3724. doi: 10.3390/nu14183724. PMID 36145099